CLINICAL TRIAL: NCT03935386
Title: A Prospective Randomized Clinical Trial Comparing Multi-layer Bandage Compression Therapy With and Without a Biologically Active Human Skin Allograft for the Treatment of Chronic Venous Leg Ulcers
Brief Title: Standard Compression Therapy With/Without Application of Skin Allograft (Theraskin) for Venous Leg Ulcer Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Solsys Medical LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soluble Inova
Record Dates: First submitted 2016-11-04; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Chronic Venous Hypertension With Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Compression (Active Comparator): Standard multi-layer compression dressing with no graft or biologic material added
  Interventions: Procedure: Standard Multi-layered Compression dressing
- Standard Compression with application of human allograft (Active Comparator): standard compression with application of a cryopreserved skin allograft (TheraSkin)
  Interventions: Procedure: Standard Multi-layered Compression dressing with a cryopreserved skin allograft (TheraSkin)

INTERVENTIONS:
Procedure: Standard Multi-layered Compression dressing — Compression therapy with a multi-layered compression dressing for the treatment of venous leg ulceration
  Arms: Standard Compression
Procedure: Standard Multi-layered Compression dressing with a cryopreserved skin allograft (TheraSkin) — Application of a cryopreserved skin allograft (TheraSkin) beneath compression therapy with a multi-layered compression dressing.
  Arms: Standard Compression with application of human allograft

SUMMARY:
This study will compare the efficacy of using standard compression therapy for treatment of chronic venous leg ulcers vs. the standard compression therapy with the additional use of the application of a human allograft (Theraskin)

DETAILED DESCRIPTION:
Given the propensity for venous leg ulcers to become refractory, long standing wounds, incorporating active biologic grafts into the standard compression therapy, may prove to accelerate wound healing. The two treatments to be compared in this study are both commonly used for the treatment of venous leg ulcers. Compression therapy has long been the standard for the treatment of venous leg ulcers. Standard Compression therapy consists of wound debridement, application of non adherent dressings and a three or four layer compression dressing. (PROFORE Multi-Layer Compression Bandage System) TheraSkin is a split thickness skin graft harvested within 24 hours postmortem, from an organ donor who has cleared the standard safety screenings. It is classified by the FDA as a donated tissue. Once harvested, the graft is sanitized according to FDA specifications, and cryopreserved, until it is delivered to the clinic for application to the foot ulcer. It is also a widely used treatment for diabetic foot ulcers. TREATMENT RATIONALE FOR THIS STUDY Chronic wounds of the lower extremities affect a substantial proportion of the population. Venous leg ulcers (VLUs) account for up to 90% of lower extremity wounds. The standard of care for treatment of VLU's in wound centers in the United States is Standard Compression therapy as described above, which may be combined with biologic graft materials applied to the wound bed. This study may assist physicians who treat VLU's by comparing efficacy and costs of two common treatments for VLU's in a prospective randomized clinical trial. The investigation will be a head-to-head study comparing widely used human skin allograft (Theraskin) along with Standard Compression Therapy vs Standard Compression Therapy alone. There is no randomized, prospective data comparing these two options in the treatment of VLU. Compression is superior to no compression and increases VLU healing rates. It is currently the mainstay of treatment for venous ulcers of the lower extremities. It is important to consider the underlying pathophysiology of these wounds. A history of deep vein thrombosis is regarded as a predisposing factor to venous insufficiency, and hence venous ulceration. Venous insufficiency is associated with increased hydrostatic pressure in the veins of the leg (Moffatt 207). External compression attempts to reverse this and aids venous return

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria: Subjects are required to meet all of the following criteria for enrollment into the study and subsequent randomization.

1. Adult patients with venous leg ulcer(s) >1 month.
2. A signed and dated informed consent form.
3. Subject is able to comply with instructions and scheduled visits, not confined to bed,.
4. Ulcer surface area >2cm2 but not >10cm in any dimension. The total not to exceed 18cm2
5. ABPI >.8, Doppler ultrasound (biphasic or triphasic waveforms) consistent with adequate blood flow to the affected extremity, as determined by the Investigator.
6. There is a minimum 2 cm margin between the qualifying study ulcer and any other ulcers on the specified leg, post-debridement) Note: If the subject has more than one qualifying VLU, the ulcer designated as the study ulcer will be at the discretion of the Investigator..
7. Casual smoker not exceeding one pack per week -

Exclusion Criteria:Exclusion Criteria: Subjects meeting any of the following criteria will be excluded from enrollment and subsequent randomization.

1. Patients with ABPI <0.7.
2. Clinical signs of infection requiring treatment. (Subjects with wound infection at the screening visit may be treated and re-screened for participation in the study after resolution of the infection).
3. Taking systemic antibiotics, steroids or immunosuppressive drugs.
4. History of poor compliance.
5. Bedridden.
6. Arterial or mixed etiology ulcers.
7. Severe diabetic peripheral neuropathy.
8. DVT in the last month.
9. Participation in another clinical investigations in the month prior to recruitment.
10. Poorly controlled hypertension.
11. Coronary artery disease.
12. Malignancy, respiratory or cardiac failure.
13. Autoimmune disease.
14. Liver (elevated enzymes)or kidney disease (elevated serum creatinine).
15. Gangrene of the affected limb.
16. Subject has suspected or confirmed signs/symptoms of gangrene or 5 wound infection on any part of the affected limb.
17. Subject has a history of hypersensitivity to any of the material used in the compression dressing
18. Subject has a history of hypersensitivity to any of the antibiotics or preservation agents listed in the TheraSkin Instructions for Use.
19. Subject was previously treated under this clinical study protocol.
20. Cytostatic therapy within the 12 months prior to randomization, dialysis, radiation therapy to the foot, vascular surgery, angioplasty or thrombolysis).
21. Subject has osteomyelitis (If the Investigator suspects the presence of osteomyelitis, the diagnosis must be confirmed by plain film Xray.)
22. Subject has a history of bone cancer or metastatic disease on the affected limb, radiation therapy to the foot or has had chemotherapy within the 12 months prior to randomization.
23. Subject has been treated with wound dressings that include growth factors, engineered tissues, or skin substitutes (e.g., Regranex®, Dermagraft®, Apligraf®, TheraSkin®, GraftJacket®, OASIS®, Primatrix®, Matristem®, etc.) within 30 days of randomization.
24. Subject has a history of or any of the following current illnesses or conditions (other than diabetes) that would compromise the safety of the subject, or the normal wound healing process:

    1. End-stage renal disease
    2. Immunosuppression
    3. Severe malnutrition
    4. Liver disease
    5. Aplastic anemia
    6. Scleroderma
    7. Acquired immune deficiency syndrome (AIDS) or HIV positive
    8. Connective tissue disorder
    9. Exacerbation of sickle cell anemia
25. Subject is an employee or relative of any member of the Investigational site or the Sponsor.
26. Subject is diabetic, HbA1c not to exceed 10% at time of enrollment.
27. COPD -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Rate of wound healing, percentage of wounds that close, and change in wound size in subjects with venous leg ulcers treated with compression therapy with or without a cryopreserved skin allograft (TheraSkin) | Enrollment and data analysis is anticipated to require approximately 3 years.
  Monitor changes in wound healing rate, percentage of wounds that close, and changes in wound size associated with two cohorts (multi-layered compression therapy vs. multi-layered compression therapy used in conjunction with a cryopreserved skin allograft.
Determine the number and severity of adverse events associated with the two treatment cohorts -- standardized multi-layered compression therapy and the same therapy with a cryopreserved skin allograft added. | Enrollment and data analysis is anticipated to require approximately 3 years.
  Measure the frequency and severity of adverse events associated with each treatment cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Garrett, DPM, Principal Investigator — Inova Hospital Wound Care Center
Locations (1):
- Inova Fairfax Hospital, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes